CLINICAL TRIAL: NCT01592825
Title: PiA Trial: a Cross-sectional, Multicenter, Consecutive Cohort Evaluating the Distribution of uPA/PAI-1 Versus St. Gallen Algorithm in >1000 Prospectively Included Patients
Brief Title: PiA: Prognosis Used Every Day for Patients With Operable Breast Cancer - Comparison of Invasion Factors uPA/PAI-1 With Other Prognostic Factors
Acronym: PiA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Eva Johanna Kantelhardt, Dr. med. E. Kantelhardt, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: GYN_Halle_01
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Prognostic factor; uPA/PA-1; cohort
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor specimen frozen Tumor specimen formalin fixed
Oversight: Data Monitoring Committee: No

SUMMARY:
The improvement of the healing rates for breast cancer is based to an important part on the consistent use of so-called adjuvant ("supporting ") medicamentous therapies, including chemotherapy. However this success has a price due to still inaccurate knowledge of the individual risk of relapse: a high number of unnecessary therapies are applied (over-therapy!). The invasion factors uPA (plasminogen activator of the urokinase type) and PAI-1 (uPA inhibitor) were described extensively as strong and independent prognosis factors with high clinical relevance for patients with node negative breast cancer. Compared to clinical and pathological factors (further: "traditional factors ") they show better estimation of the relapse risk leading to an avoidance of redundant adjuvant chemotherapy and may thus essentially contribute to the improvement of the quality of life in these women. In this study we aim to evaluate, how large the portion of the patients with early, operable, node negative breast cancer will be, in whom, by improved low-risk identification through uPA/PAI-1, adjuvant chemotherapy can be omitted.

DETAILED DESCRIPTION:
The determination of the prognostic factors uPA/PAI-1 (further: "biological") is established and recommend by recent guidelines. However, so far data can only show their independent and strong prognostic influence. The absolute proportion of patients, which profit from the improved risk assessment, is only estimated from old trials with different patient populations.

Depending upon assessment, the proportion of low risk patients by traditional risk assessment is 20 - 40%, by biological assessment 35 - 55% of all node negative patients. The data from investigations of historic populations are not reproducible now because of smaller tumor size at presentation due to diagnostic procedures (Screening, good public promotion).

The effectiveness and clinical relevance of the risk assessment were already confirmed for the biological prognostic factors uPA/PAI-1 in node negative breast cancer in several retrospective and prospective trials as well as in a meta-analysis. Still these biological factors (or others!) are not yet established into nationwide clinical routine in Germany. This is due to higher expenditure of this method for the primary therapy (uPA/PAI-1 is determined in the shock-frozen tissue), on the other hand due to the absence of reimbursement. Therefore presently in many centres risk estimation and associated therapy decision is done by traditional assessment.

In order to justify the higher expenditure and the additional costs by the uPA/PAI-1-determination, not only the clear proof of the advantage for the individual patient, but also the estimation of the extent of this advantage in all applicable patients is necessary.

A first goal of this project is to compare the respective proportion of patients allocated as high- or low-risk by means of biological and also traditional prognosis factors in a defined consecutive patient cohort. The determination of uPA/PAI-1 should be established as standard procedure in the future.

So far, the question discussed above referred mainly to patients with node negative breast cancer. In this group, the largest effect in saving chemotherapy is to be expected. Due to previous results we assume that also in node positive patients adjuvant chemotherapy may be saved in sub-group because of very small risk of recurrence. Therefore the determination of uPA/PAI-1 for this group of patients will also be done at the end of this study.

A second goal of this project is it to collect data for risk assessment in node positive patients to be able to offer assistance in the future to perhaps give a better estimation of the individual risk of recurrence.

Practically fresh frozen tissue will be taken, shock-frozen and stored from all consecutive patients operated in the five participating hospitals. The determination of uPA/PAI-1 will be performed in the research laboratory of department of Gynaecology at the University Hospital in Halle (Saale).

A third goal is it to provide biological risk assessment by giving results of uPA/PAI-1 testing promptly to participating node negative patients. This information will be crucial in their decision for or against chemotherapy.

Amendment 2 from June 12, 2012 (Steering committee E Kantelhardt, M Vetter, Ch Thomssen)

A) Established prognostic factors (RNA level) will be evaluated in the context of uPA/PAI-1 and immunohistochemistry markers on samples from the frozen and FFPE tissue. The list of genes is submitted to the Ethics sommittee.

B) Eplorative analysis of these factors concerning response to therapy will be done.

C) Follow-up information will be collected after a minimum observation time of 2.5 years for all patients (in October 2013).

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed breast cancer
* no metastasis detected
* operation for breast cancer
* female patient
* unilateral breast cancer
* informed consent given
* age min. 18 yrs.

Exclusion Criteria:

* metastasis of breast cancer
* bilateral breast cancer
* other cancer within the last 5yrs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed, operable breast cancer without metastasis.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 2.5 years minimum observation time
  All patients will be followed after a minimum observation time of 2.5 years.

SECONDARY OUTCOMES:
Overall survival | 2.5 years
  All patients will be followed after a minimum observation time of 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eva J Kantelhardt, MD, Principal Investigator — Gynecology Martin Luther Univ Halle/Germany

REFERENCES:
- [Derived] Engel J, Wieder V, Bauer M, Kaufhold S, Stuckrath K, Wilke J, Hanf V, Uleer C, Lantzsch T, Peschel S, John J, Pohler M, Weigert E, Burrig KF, Buchmann J, Santos P, Kantelhardt EJ, Thomssen C, Vetter M. Prognostic and predictive impact of NOTCH1 in early breast cancer. Breast Cancer Res Treat. 2025 Jan;209(1):27-38. doi: 10.1007/s10549-024-07444-1. Epub 2024 Aug 17. PMID 39153127
- [Derived] Breunig C, Erdem N, Bott A, Greiwe JF, Reinz E, Bernhardt S, Giacomelli C, Wachter A, Kanthelhardt EJ, Beissbarth T, Vetter M, Wiemann S. TGFbeta1 regulates HGF-induced cell migration and hepatocyte growth factor receptor MET expression via C-ets-1 and miR-128-3p in basal-like breast cancer. Mol Oncol. 2018 Sep;12(9):1447-1463. doi: 10.1002/1878-0261.12355. Epub 2018 Jul 30. PMID 30004628
- [Derived] Bernhardt S, Bayerlova M, Vetter M, Wachter A, Mitra D, Hanf V, Lantzsch T, Uleer C, Peschel S, John J, Buchmann J, Weigert E, Burrig KF, Thomssen C, Korf U, Beissbarth T, Wiemann S, Kantelhardt EJ. Proteomic profiling of breast cancer metabolism identifies SHMT2 and ASCT2 as prognostic factors. Breast Cancer Res. 2017 Oct 11;19(1):112. doi: 10.1186/s13058-017-0905-7. PMID 29020998